CLINICAL TRIAL: NCT02990182
Title: Complementary Study of the Duration of Post-vaccination Against Yellow Fever Immunity in Children
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oswaldo Cruz Foundation (Other)
Responsible Party: Principal Investigator, Olindo de Assis Martins Filho, PhD, Oswaldo Cruz Foundation
Other Study IDs: CPqRR - M 02
Record Dates: First submitted 2015-09-01; First posted 2016-12-13 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Yellow Fever
Keywords: Yellow Fever Vaccine; Immunity, Humoral; Immunity, Cellular; children
MeSH Terms: conditions — Yellow Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood and plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
In a previous study by the researchers' group, the researchers' investigate the duration of yellow fever post-vaccination immunity in vaccinated children between 9 and 23 months of age. However, in this study, samples of children in the pre-vaccine period, also known as unvaccinated children samples (NV) have not been investigated. It is believed that to seek evidence about the immune status in the medium and long term after vaccination against yellow fever is necessary to investigate paired samples of children not vaccinated (NV), with re-evaluation 30-45 days after primary vaccination. The proposed study is to consolidate aspects of humoral (neutralizing antibodies) and cellular (phenotypic and functional parameters of T cells and memory B) by means of complementary longitudinal investigation children, 9-23 months old, unvaccinated (NV) and 30-45 days after primary vaccination.

DETAILED DESCRIPTION:
A sample of 60 children aged 9 to 23 months paired in the pre-vaccine period (NV) and 30-45 post-primary vaccination days will be selected at health facilities in the metropolitan region of Belo Horizonte.

Children whose mothers consent to participate in research, have collected blood and elements of past medical history recorded. Analyses of humoral and cellular biomarkers will be used in a comparative study with other post-vaccination periods previously analyzed in children during the first phase in study funded by the Ministry of Health.

specific objectives:

1. Estimate and compare the proportion of positivity and the geometric mean plasma titers of neutralizing antibodies against yellow fever;
2. Assess lymphocyte frequency T and B memory induced in vitro by the vaccine antigen 17DD substrains, and...
3. Quantify the lymphocytes T CD8 + producers of intracytoplasmic cytokines induced in vitro by the vaccine antigen 17DD substrains in unvaccinated children and primed aged between 9 and 23 months, categorized according to the vaccination time 30-45 days.

ELIGIBILITY:
Inclusion Criteria:

Will be eligible for the study:

* children 9-23 months of age;
* both sexes;
* children who will be vaccinated against yellow fever, whose parents or guardians sign the consent form.

Exclusion Criteria:

* children who received another vaccine within 30 days before or after the yellow fever vaccine;
* children which have permanent or temporary immunosuppression, including those treated with corticosteroids at doses higher than 2 mg / kg, and those with disease autoimmune diseases, transient or permanent immunosuppression induced diseases (cancer, AIDS, etc.) or treatment (immunosuppressive drugs, radiotherapy, etc.). Corticosteroids (such as prednisone, dexamethasone) for less than two weeks, or by inhalation or topical use, do not indicate exclusion from the study, but must be registered in the questionnaire (Annex II);
* children with hemoglobinopathies;
* children with a history of blood transfusion or treatment with hyperimmune serum up to 90 days prior to blood collection.

Ages: 9 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study provides immunoassays paired before and after anti-yellow fever vaccination in children of both sexes, of any color, class or social group. This will be necessary 60 paired samples (pre-vaccine period and 30-45 days after primary vaccination) of children aged 9 to 23 months, living in areas where YF vaccine makes up the basic immunization calendar and will receive the vaccine in the routine of UBRs in the first two years of life. This study will be conducted with samples collected from children living in Ribeirão das Neves - Minas Gerais. It will be collected 7 mL of whole blood collected in Heparin Sodium. It will be allowed to make two attempts to collect only. These samples will be used for the realization of the humoral and cellular immunity study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2017-04 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Quantification of Humoral and cellular immunity after first yellow fever vaccination | Time 0 (immediately before) and Time 1 (30-45 days after) primary vaccination against yellow fever
  Consolidating aspects of humoral (quantification of neutralizing antibodies - >2.log10IU/mL) and cellular (Percentege of phenotypic and functional parameters of T cells and B memory) through a complementary longitudinal investigation in children aged 9 to 23 month old unvaccinated and 30-45 days after first vaccination .

SECONDARY OUTCOMES:
Quantification of titers of neutralizing antibodies in plasma samples | Time 0 (immediately before) and Time 1 (30-45 days after) primary vaccination against yellow fever
  Quantify the titers of neutralizing antibodies against yellow fever immediately before and 30-45 days after primary vaccination against yellow fever in children 9-23 months of age without yellow fever vaccination history.
Evaluate the frequency (percentage) of T cells and B memory induced in vitro by the vaccine antigen 17DD | Time 0 (immediately before) and Time 1 (30-45 days after) primary vaccination against yellow fever
  Evaluate the frequency (percentage) of T cells and B memory induced in vitro by the vaccine antigen 17DD immediately before and 30-45 days after primary vaccination against yellow fever in children 9-23 months old with no vaccination history against yellow fever.
Evaluate the frequency (percentage) of T and B cells expressing intracytoplasmic cytokines in vitro induced by the vaccine antigen 17DD | Time 0 (immediately before) and Time 1 (30-45 days after) primary vaccination against yellow fever
  Evaluate the frequency (percentage) of T and B cells expressing intracytoplasmic cytokines (gama interferon; IL-5, alfa-TNF) CD8 + T lymphocytes, in vitro induced by the vaccine antigen 17DD immediately before and 30-45 days after primary vaccination against yellow fever, in children 9-23 months of age without yellow fever vaccination history.

CONTACTS AND LOCATIONS:
Overall Officials: Olindo A Martins-Filho, PhD, Principal Investigator — Centro de Pesquisas René Rachou
Locations (1):
- Centro de Pesquisas René Rachou, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] Vasconcelos PF. [Yellow Fever]. Rev Soc Bras Med Trop. 2003 Mar-Apr;36(2):275-93. doi: 10.1590/s0037-86822003000200012. Epub 2003 Jun 10. Portuguese. PMID 12806465
- [Result] ANDERSON CR, GAST-GALVIS A. Immunity to yellow fever five years after vaccination. Am J Hyg. 1947 May;45(3):302-4. doi: 10.1093/oxfordjournals.aje.a119138. No abstract available. PMID 20240017
- [Result] Belmusto-Worn VE, Sanchez JL, McCarthy K, Nichols R, Bautista CT, Magill AJ, Pastor-Cauna G, Echevarria C, Laguna-Torres VA, Samame BK, Baldeon ME, Burans JP, Olson JG, Bedford P, Kitchener S, Monath TP. Randomized, double-blind, phase III, pivotal field trial of the comparative immunogenicity, safety, and tolerability of two yellow fever 17D vaccines (Arilvax and YF-VAX) in healthy infants and children in Peru. Am J Trop Med Hyg. 2005 Feb;72(2):189-97. PMID 15741556
- [Result] Camacho LA, Freire Mda S, Leal Mda L, Aguiar SG, Nascimento JP, Iguchi T, Lozana Jde A, Farias RH; Collaborative Group for the Study of Yellow Fever Vaccines. Immunogenicity of WHO-17D and Brazilian 17DD yellow fever vaccines: a randomized trial. Rev Saude Publica. 2004 Oct;38(5):671-8. doi: 10.1590/s0034-89102004000500009. Epub 2004 Oct 18. PMID 15499438
- [Result] Collaborative Group for Studies with Yellow Fever; Camacho LAB. Immunogenicity of 17DD and WHO 17D -213/77 Yellow Fever Vaccines in Children less than 2 years old: a randomized, double-blind study. In: 5th World Congress of the World Society fo Pediatric Infectious Diseases, 2007, Bangkok, Tailandia. Book of Abstracts, 2007.
- [Result] Collaborative Group for Studies with Yellow Fever Vaccine. Randomized, double-blind, multicenter study of the immunogenicity and reactogenicity of 17DD and WHO 17D-213/77 yellow fever vaccines in children: implications for the Brazilian National Immunization Program. Vaccine. 2007 Apr 20;25(16):3118-23. doi: 10.1016/j.vaccine.2007.01.053. Epub 2007 Jan 22. PMID 17316925
- [Result] FOX JP, FONSECA DA CUNHA J, KOSSOBUDZKI SL. Additional observations on the duration of humoral immunity following vaccination with the 17D strain of yellow fever virus. Am J Hyg. 1948 Jan;47(1):64-70. doi: 10.1093/oxfordjournals.aje.a119186. No abstract available. PMID 18921440
- [Result] Hepburn MJ, Kortepeter MG, Pittman PR, Boudreau EF, Mangiafico JA, Buck PA, Norris SL, Anderson EL. Neutralizing antibody response to booster vaccination with the 17d yellow fever vaccine. Vaccine. 2006 Apr 5;24(15):2843-9. doi: 10.1016/j.vaccine.2005.12.055. Epub 2006 Jan 18. PMID 16494976
- [Result] Monath TP, Cetron MS & Teuwen DE. Yellow fever vaccine. In Plotkin SA, Orenstein WA & Offit P. Organizadores. Vaccine. Philadelphia. Saunders Elsevier 2008. p. 959-1056.
- [Result] Niedrig M, Lademann M, Emmerich P, Lafrenz M. Assessment of IgG antibodies against yellow fever virus after vaccination with 17D by different assays: neutralization test, haemagglutination inhibition test, immunofluorescence assay and ELISA. Trop Med Int Health. 1999 Dec;4(12):867-71. doi: 10.1046/j.1365-3156.1999.00496.x. PMID 10632996
- [Result] Poland JD, Calisher CH, Monath TP, Downs WG, Murphy K. Persistence of neutralizing antibody 30-35 years after immunization with 17D yellow fever vaccine. Bull World Health Organ. 1981;59(6):895-900. PMID 6978196
- See also: World Health Organization.International health regulations (2005) — http://www.who.int/
- See also: Ministério da Saúde. Secretaria de Vigilância em Saúde. Departamento de Vigilância Epidemiológica. Guia de Vigilância Epidemiológica. 6ª edição. Série A. Normas e Manuais Técnicos. Brasília - DF, 2005. — http://portalsaude.saude.gov.br/